CLINICAL TRIAL: NCT05521074
Title: Transcranial Direct Current Stimulation Potentiation of Fear Extinction in OCD: Towards Rational Design of Combination Therapies
Brief Title: Transcranial Direct Current Stimulation Potentiation of Fear Extinction in OCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Foundation for OCD Research (Unknown)
Responsible Party: Principal Investigator, Joan A Camprodon, MD MPH PhD, PI of IRB Protocol, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2022P001065
Record Dates: First submitted 2022-08-26; First posted 2022-08-30 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Obsessive-Compulsive Disorder; OCD; Fear extinction; tDCS; transcranial Direct Current Stimulation; Randomized controlled trial; Fear conditioning
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- Active tDCS administered before extinction phase (Experimental): The investigators will stimulate using 2mA of direct current during 20 min before the extinction phase of the fear conditioning and extinction paradigm.
  Interventions: Device: Active tDCS
- Active tDCS administered during extinction phase (Experimental): The investigators will stimulate using 2mA of direct current during 20 min during the extinction phase of the fear conditioning and extinction paradigm.
  Interventions: Device: Active tDCS
- Active tDCS administered after extinction phase (Experimental): The investigators will stimulate using 2mA of direct current during 20 min after the extinction phase of the fear conditioning and extinction paradigm.
  Interventions: Device: Active tDCS
- Sham tDCS (Sham Comparator): Sham will consist of a ramp up and down of activity (from 0 to 2mA and back to 0mA) in the first 30sec and again in the last 30 sec of the 20min stimulation period (which will occur before/during/after the extinction phase). No active tDCS will occur.
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Active tDCS — The investigators will use commercially available tDCS equipment (Neuroelectrics©, Barcelona, Spain). The cathode will be placed over the pre-SMA using the 10-20 EEG system and the anode will be on the right deltoid.
  Arms: Active tDCS administered after extinction phase; Active tDCS administered before extinction phase; Active tDCS administered during extinction phase
Device: Sham tDCS — The investigators will use commercially available tDCS equipment (Neuroelectrics©, Barcelona, Spain). The cathode will be placed over the pre-SMA using the 10-20 EEG system and the anode will be on the right deltoid. tDCS will not be active in this condition.
  Arms: Sham tDCS

SUMMARY:
The investigators want to learn more about how human beings learn not to fear and the impact of changing the fear network in the brain using transcranial Direct Current Stimulation (tDCS) in individuals with obsessive compulsive disorder (OCD). The investigators hope this study will help us understand how future treatments can help patients with OCD better control unwanted fear.

DETAILED DESCRIPTION:
To address this question behaviorally and biologically, the investigators will use a, 2-day fear extinction paradigm while measuring behavioral psychophysiology (skin conductance response [SCR]) and neurophysiology (electroencephalography [EEG]). On Day 1 participants will undergo 1) habituation, 2) fear conditioning, and 3) extinction learning. On Day 2 they will undergo 4) extinction recall, and 5) reinstatement. SCR and EEG will be measured in both sessions. The investigators propose to investigate whether inhibitory tDCS to the pre-SMA before, during, or after fear extinction significantly 1) enhances the recall of extinction learning and 2) reduces fronto-medial theta power during extinction recall. Participants will be randomized to one of the following four conditions: active tDCS before, during, or after extinction learning, or sham tDCS. The fear extinction paradigm serves as a proxy of exposure-based CBT for OCD. Defining the combination protocol that optimally and significantly increases extinction recall behaviorally (psychophysiology) in OCD, will have critical implications for the mechanistically informed development of tDCS-augmented CBT for OCD. EEG measures will provide a response biomarker to characterize target engagement neurophysiologically. This is particularly relevant given EEG's ease of use, relatively low cost, and potential for greater translation to the clinic. Also, the higher signal-to-noise ratio (SNR) of EEG compared to SCR is a strength. Taken together, these data should reveal treatment targets, define optimal therapeutic protocols, and provide the foundation for a future clinical trial to test the synergistic efficacy of combined tDCS-CBT for OCD.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English, willing to provide informed consent, and willing to comply with the study protocol
* Primary OCD that causes at least moderate distress and/or impairment (Y-BOCS total score ≥ 16)
* Comfortable and capable of using a computer and completing computerized tasks

Exclusion Criteria:

* History of head injury resulting in prolonged (i.e., >1h) loss of consciousness and/or neurological sequelae; history of stroke; signs of increased intracranial pressure; prior neurosurgical procedure (e.g., DBS, aneurysm clips)
* Contraindications to participate in tDCS including: metallic implants in head or neck; ventriculoperitoneal (VP) shunts; pacemakers; pregnancy; epilepsy.
* Current or history of neurologic or psychiatric disease (e.g., mental retardation, dementia, brain damage, or other cognitive impairment) that would interfere with ability to participate in the study
* Impaired (or uncorrected) vision that would interfere with participation.
* Current clinically significant suicidality that requires psychiatric hospitalization, as indicated by clinical judgment.
* Current substance use disorder (within the past 12 months)
* Lifetime manic episode or psychosis
* Documented resistance to 4 or more valid pharmacological trials and previous treatment with ≥12 sessions of cognitive behavioral therapy for OCD with no response (or worsening symptoms)
* Use of most psychotropic medications (e.g., SSRIs and atypical antipsychotics) will be allowed. However, use of benzodiazepines within 2 weeks prior to the study is exclusionary (and participants will be asked to refrain from use of such medications during the study as they may interfere with the fear extinction paradigm).
* Unable to obtain low enough impedance values to ensure safe and effective application of tDCS/EEG.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Difference in skin conductance response (SCR) to the conditioned stimulus (CS+) versus the unconditioned stimulus (CS-) between tDCS conditions during extinction recall | Extinction Recall Phase (Day 2)
  Higher skin conductance (microSiemens) indicates greater fear intensity.
Difference in frontomedial theta power (EEG) to the conditioned stimulus (CS+) versus the unconditioned stimulus (CS-) between tDCS conditions during extinction recall | Extinction Recall Phase (Day 2)
  Greater reduction of frontomedial theta power (microvolts) indicates stronger extinction recall.

CONTACTS AND LOCATIONS:
Overall Officials: Joan Camprodon, MD, MPH, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
The investigators do not have specific plans to share individual participant data in order to preserve the confidentiality of our participants. Any data that is shared would only be done so after executing a formal Data Use Agreement from Massachusetts General Hospital.

REFERENCES:
- See also: Eligibility Interest Form — https://redcap.link/ocdfearstudy_prescreen